CLINICAL TRIAL: NCT01468623
Title: A Prospective, Randomized, Open-label Trial Comparing OnDose® AUC Optimized 5-FU Based Administration Versus Standard Body Surface Area (BSA) Dosing in Metastatic Colorectal Cancer Patients (mCRC) Treated With mFOLFOX6
Brief Title: Study Comparing Optimized 5-FU Dosing and Standard Dosing in Metastatic Colorectal Cancer Patients Treated With mFOLFOX6
Acronym: PROFUSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment.
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROFUSE-2011
Record Dates: First submitted 2011-11-01; First posted 2011-11-09 (Estimated); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer, Metastatic
Keywords: Colorectal cancer, metastatic; FOLFOX6; 5-FU; First line; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OnDose® (Experimental): Patients will receive FOLFOX6 with or without bevacizumab (Avastin). Patients' 5-FU dose will be optimized by measuring the Area Under the Curve (AUC) of 5-FU by the commercially available OnDose® assay and their dose for subsequent cycles adjusted following a pre-established dose adjustment algorithm.
  Interventions: Other: Pharmacokinetic 5-FU dose adjustment using OnDose® assay
- Body Surface Area (BSA) (Active Comparator): Patients will receive FOLFOX6 with or without bevacizumab (Avastin). Patients will receive 5-FU based on traditional BSA calculation and their dose adjusted based on standard clinical practice. OnDose® AUC measurements will be performed for this arm but will not be used for dose adjustment.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Pharmacokinetic 5-FU dose adjustment using OnDose® assay — OnDose is a commercially available assay to measure concentration of 5-FU exposure.
  Other Names: OnDose®
  Arms: OnDose®
Other: Standard of care — Patients' dose of 5-FU will be based on Body Surface Area (BSA).
  Arms: Body Surface Area (BSA)

SUMMARY:
The purpose of this study is to compare OnDose® based pharmacokinetic administration of 5-FU versus standard Body Surface Area (BSA) based administration of 5-FU in patients with metastatic colorectal cancer treated with mFOLFOX6, with or without bevacizumab, to determine if the use of OnDose® achieves an improvement in the Overall Response Rate (ORR) relative to BSA dosing response.

ELIGIBILITY:
Selection Criteria:

* Patients with histologically confirmed metastatic colorectal cancer
* No prior chemotherapy for the treatment of metastatic colorectal cancer
* At least one measurable lesion by CT or MRI of ≥ 20 mm (if conventional CT scan) or ≥ 10 mm (if spiral CT scan)
* ECOG Performance Status (ECOG-PS) status ≤ 2
* At least 18 years of age
* Life expectancy > 6 months
* Must be able and willing to give written informed consent
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Nursing patients are excluded. Sexually active men must also use acceptable contraceptive methods (abstinence, condom).
* ANC count greater than or equal to 1,500/ mm³
* Platelets greater than or equal to 100,000/ mm³
* Serum creatinine less than or equal to 2x upper limit of normal (normal range (male): 97-137 mL/min; (female): 88-128 mL/min)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3x the upper limit of normal (≤ 5.0 x ULN is acceptable if liver has tumor involvement) (ALT normal range: < 41 iu/L (male), < 31 iu/L (female); AST normal range: < 37 iu/L (male), < 31 iu/L (female)).
* Prothrombin Time (PT), activated partial thromboplastin time (aPTT) and INR ≤ 1.5 x ULN (INR normal range: 0.8-1.2) or in the therapeutic range if on anticoagulation.
* Hemoglobin greater than or equal to 9 gm/dl (may be corrected by transfusion prior to 5-FU treatment with investigator approval).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Abebe Haregewoin, MD, PhD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (58):
- United States (58):
  - Birmingham, Alabama
  - Corona, California
  - Fountain Valley, California
  - La Jolla, California
  - Modesto, California
  - Rancho Cucamonga, California
  - Riverside, California
  - Santa Rosa, California
  - Washington D.C., District of Columbia
  - Merritt Island, Florida
  - Ocala, Florida
  - Titusville, Florida
  - Viera, Florida
  - Albany, Georgia
  - Chicago, Illinois
  - Crystal Lake, Illinois
  - Galesburg, Illinois
  - Grayslake, Illinois
  - Highland Park, Illinois
  - Lake Forest, Illinois
  - Libertyville, Illinois
  - Niles, Illinois
  - Skokie, Illinois
  - Munster, Indiana
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Metairie, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Farmington Hills, Michigan
  - Great Falls, Montana
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - Johnson City, New York
  - Greensboro, North Carolina
  - Fargo, North Dakota
  - Minot, North Dakota
  - Canton, Ohio
  - Columbus, Ohio
  - Bend, Oregon
  - Drexel Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Crossville, Tennessee
  - Huntsville, Tennessee
  - Bedford, Texas
  - Garland, Texas
  - Grapevine, Texas
  - Kerrville, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Waco, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Newport News, Virginia
  - Edmonds, Washington
  - Seattle, Washington